CLINICAL TRIAL: NCT02253602
Title: Innovative MRI Techniques to Improve Treatment Stratification of Patients With Esophageal Cancer: an Optimization and Pilot Study
Brief Title: Innovative MRI Techniques to Improve Treatment Stratification of Patients With Esophageal Cancer
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL48757.018.14
Record Dates: First submitted 2014-09-04; First posted 2014-10-01 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal Neoplasms; Lymph Nodes; USPIO; Magnetic Resonance Imaging
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Ferrosoferric Oxide; ferumoxtran-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ferumoxytol Dose optimization (Experimental): We will assess three different dose levels of Ferumoxytol (4 mg/kg, 6 mg/kg, 8 mg/kg).
  Images will be acquired at baseline (before Ferumoxytol administration), during injection of Ferumoxytol and 24, 48 and 72 hours after Ferumoxytol administration to identify the optimal moment of scanning.To assess whether USPIOs are sufficiently cleared within 12 weeks from lymph nodes, the MRI scans will be repeated in all six volunteers at 12 weeks after Ferumoxytol administration. Thus, volunteers will undergo an MRI scan for five times. Ferumoxytol is administered only once
  Interventions: Drug: Ferumoxytol
- Before Surgery (Experimental): Twenty patients will be measured directly before surgery. Patients will be measured at baseline, during injection of Ferumoxytol and 24, 48 or 72 hours after Ferumoxytol administration, depending on the results of the dose optimization study. MR parameters will be correlated with pathology data.
  Interventions: Drug: Ferumoxytol
- Before Neoadjucant therapy (Experimental): Ten patients will be measured before start of neoadjuvant chemoradiation. Patients will be measured at baseline, during injection of Ferumoxytol and 24, 48 or 72 hours after Ferumoxytol administration, based on the dose optimization study. MR parameters will be correlated with pathology data.
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — maximum rate of administration 1 ml/sec
  Other Names: USPIO; Rienso

SUMMARY:
The current standard treatment of resectable esophageal cancer consists of neoadjuvant chemoradiation followed by resection. However, some patients develop recurrent disease despite chemoradiation and additional (systemic) treatment might have been indicated. Other patients show a (nearly) complete response after chemoradiation and could possibly have been treated with a less extensive treatment regimen. In patients without a threatened circumferential resection margin (CRM) and lymph node metastases chemoradiotherapy could possibly be omitted.

Better stratification of patients with esophageal cancer is therefore urgently needed. Functional magnetic resonance imaging techniques (MRI) can provide in vivo, quantitative information on tumor biology and may prove to be a useful non-invasive tool for this purpose. In this project, ultra-small superparamagnetic particles of iron oxide (USPIO) enhanced MRI using ferumoxytol (Rienso®), diffusion weighted MRI (DWI) and T2* MRI will be developed, both in terms of improvement of acquisition and data processing techniques.

DETAILED DESCRIPTION:
The outcome of esophageal cancer is poor, with an overall 5-year survival rate of 10% worldwide. In resectable esophageal cancer, outcome can be improved by multimodality treatment. The current standard treatment of resectable esophageal cancer consists of neoadjuvant chemoradiation followed by resection. In the Netherlands, the preferred chemoradiation regimen consists of carboplatin plus paclitaxel with concurrent radiotherapy in 23 fractions of 1.8 Gray.1 In a meta-analysis the benefit of chemoradiation over surgery alone for both adenocarcinoma and squamous cell carcinoma has been shown.2 However, not all patients benefit from this preoperative treatment regimen. Some patients develop recurrent disease despite chemoradiation and additional (systemic) treatment might have been indicated. In contrast, in other patients a (nearly) complete response is observed after chemoradiation and those patients could possibly have been treated with a less extensive treatment regimen. Furthermore, in patients without a threatened circumferential resection margin (CRM) and lymph node metastases chemoradiotherapy could possibly be omitted, reducing patients' risk for complications and unnecessary, expensive treatment. Thus, stratification of patients with esophageal cancer is urgently needed. Functional magnetic resonance imaging techniques (MRI) can provide in vivo, quantitative information on tumor biology and may prove to be a useful non-invasive tool for this purpose. In this project, ultra-small superparamagnetic particles of iron oxide (USPIO) enhanced MRI using ferumoxytol (Rienso®), diffusion weighted MRI (DWI) and T2* MRI will be developed, both in terms of improvement of acquisition and data processing techniques. For patients with esophageal cancer, the proposed acquisition techniques and data processing have not been performed before.

Objectives of the study

1. To determine the optimal acquisition technique for USPIO enhanced MRI and DWI and T2* MRI of esophageal cancer in terms of signal-to-noise ratio, time resolution and spatial resolution.
2. To determine the optimal data processing approach for USPIO enhanced MRI, DWI and T2* MRI of esophageal cancer.
3. To explore the correlation between lymph node involvement on USPIO enhanced MRI in relation to results obtained at pathological examination.
4. To explore the correlation of DWI and T2* MRI of esophageal cancer in relation to stromal involvement and markers of hypoxia and vasculature obtained at pathological examination.
5. To explore the accuracy of MRI concerning circumferential tumor delineation compared to pathological examination.
6. To determine the feasibility to detect lymph node involvement on USPIO enhanced MRI in initial staging, prior to preoperative chemoradiation therapy.
7. To determine the correlation between lymph node involvement on pre-treatment USPIO MRI in relation to results obtained at pathology after complete treatment.

The project will be executed in four steps:

1. Optimization of acquisition and data processing techniques of USPIO MRI, DWI and T2* in five healthy volunteers to optimize field of view, number of slices, slice thickness (objectives 1 and 2).
2. Assessment of ferumoxytol dose-response with three different dose levels at three different time points in six healthy volunteers (two per dose-level) (objectives 1 and 2).
3. Using the data of (1) and (2): assessment of USPIO MRI, DWI and T2* MRI in 20 esophageal cancer patients with clinically suspect lymph nodes directly before surgery (objectives 3, 4 and 5).
4. Using the data of (1) and (2): assessment of USPIO MRI, DWI and T2* MRI in 10 esophageal cancer patients with clinically suspect lymph nodes, before initial start of the treatment (objectives 6 and 7).

For step 1 and 2 we aim to include healthy volunteers; for step 3 and 4 we aim to include patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven esophageal cancer (squamous cell carcinoma or adenocarcinoma)
* Suspected nodal involvement on EUS or CT at diagnosis.
* WHO-performance score 0-2
* Scheduled for surgery
* Written informed consent

Exclusion Criteria:

* Any psychological, familial, sociological or geographical condition potentially hampering adequate informed consent or compliance with the study protocol
* Contra-indications for MR scanning, including patients with a pacemaker, cochlear implant or neurostimulator; patients with non-MR compatible metallic implants in their eye, spine, thorax or abdomen; or a non-MR compatible aneurysm clip in their brain; patients with severe claustrophobia
* Active inflammatory diseases
* History of anaphylaxis or other hypersensitivity reactions
* History of iron overload
* History of abnormal liver function, or elevated liver enzymes (ALAT, ASAT > 3 times upper limit of normal)
* Elevated Serum Transferrin Saturation (TSAT) (>50%) or hemoglobin (>10.5mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
USPIO MRI | 24, 48 or 72 hours after USPIO administration
  For USPIO enhanced MRI the main endpoint is the change in T2 and T2* at the tumor and lymph nodes on MRI after the administration of USPIO.
DWI/IVIM MRI | 1 hour before USPIO administration
  For DWI the main endpoint is the perfusion fraction f and the diffusion coefficient D obtained by IVIM of the primary tumor.
T2* MRI | 1 hour before USPIO administration
  For T2* MRI the main endpoint is T2* of the primary tumor
Ferumoxytol dose response | 24, 48, 72 hours and 12 weeks after the administration of Ferumoxytol
  For Ferumoxytol dose evaluation the main endpoint is the change in T2 and T2* at the tumor and lymph nodes on MRI at 24, 48, 72 hours and 12 weeks after the administration of Ferumoxytol.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke WM van Laarhoven, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands